CLINICAL TRIAL: NCT04294316
Title: Evaluation of Cerebral Microcirculation Using Non-invasive Contrast-enhanced Ultrasound and Microbubbles Sonovue Administration After Clinical Cardiorespiratory Arrest
Brief Title: Enhanced-contrast Brain Ultrasound in Cardiorespiratory Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Duc Nam Nguyen, Clinical Professor, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B.U.N 143201941163
Record Dates: First submitted 2020-02-29; First posted 2020-03-04 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-02

CONDITIONS: Cardiorespiratory Arrest; Microcirculation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: ICU patients with successful resuscitation after out-hospital or in-hospital cardiorespiratory arrest who are eligible for enhanced-contrast brain ultrasound with sulphur hexafluoride microbubbles contrast Sonovue examination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonovue group (Other): ICU patients with successful resuscitation after out-hospital or in-hospital cardiorespiratory arrest who are eligible for enhanced-contrast brain ultrasound, extracranial echo-color duplex, and ocular ultrasound.
  Interventions: Diagnostic Test: Sonovue

INTERVENTIONS:
Diagnostic Test: Sonovue — Twice dose of 2.4ml of Sulphur hexafluoride microbubbles contrast Sonovue administration to evaluate brain microcirculation

SUMMARY:
Brain microcirculation alterations may be involved in comatose patients and non-survivors after cardiorespiratory arrest. For a three day-period, we investigate brain microcirculation using contrast-enhanced ultrasound with contrast Sonovue injection in patients with successful resuscitation after out-hospital or in-hospital cardiorespiratory arrest.

DETAILED DESCRIPTION:
Brain ultrasound, extracranial echo-color duplex and ocular ultrasound (IE 33, Philips Medical System, the Netherlands) are performed in the first 24 hours, at 48 hours, and at 72-96 hours after successful resuscitation after out-hospital or in-hospital cardiorespiratory arrest.

Ultrasound examinations are performed in four steps to 1) evaluate the global cerebral blood volume, 2) to estimate the presence or absence of cerebral autoregulation, and 3) to qualitatively evaluate the cerebral perfusion and microcirculation by enhanced microbubbles contrast injection 4) to qualitatively evaluate the intracranial pressure.

Before performing brain ultrasound, echocardiography (IE 33, Philips medical System, the Netherlands) is performed to evaluate the cardiac output (L/min).

First, the global cerebral blood volume (L/min) is evaluated as the sum of flow volumes of the internal carotid (ICA) and vertebral arteries (VA) extracranial arteries of both sides.The following measurements of flow velocities are taken in each artery: Peak systolic and end-diastolic velocity, time-averaged velocity (TAV), Pulsatility Index (PI). Flow volume (Q) of each artery is determined as Q = TAV x Area ((diameter of the artery /2)² x PI).

Brain ultrasound is performed via temporal windows to measure the mean flow velocities (cm/sec) of the middle cerebral arteries.

Second, the presence or absence of cerebral autoregulation is tested with the Transient hyperemic response by an ipsilateral common carotid compression one side and another during 5 seconds. Absence of cerebral autoregulation is considered if the flow velocity of the middle cerebral artery do not increase more than 10% after the compression.

Third, the brain regional microcirculation is evaluated by the microbubbles contrast injection of Sonovue. The brain parenchyma is insonated via the temporal bone windows at the depth of 10cm with the ultrasound S5 multifrequency transducer 2-5 Megahertz (MHz) probe. After optimizing the acoustic bone window, Sonovue is injected intravenously as a bolus 2.4ml followed by 10ml saline flushed. The contralateral brain is evaluated 5 minutes after the first injection of Sonovue to allow a complete evacuation of contrast microbubbles.

All real-time images are stored digitally on the hard disk as DICOM (Digital Image Communications in Medicine) images. Offline imaging analysis using a specific quantification software named QLAB10 (Philips Medical System, the Netherlands) to convert brain perfusion images into time-intensity curves (TIC) corresponding to the five different regions of interest (ROI) of brain parenchyma: anterior and posterior thalamus, lentiform nucleus, parieto-temporal and posterior white matter. Four variables were extracted from these TIC curves to qualitatively evaluate the brain microcirculation: peak intensity in dB, time to peak intensity in seconds, mean transit time in seconds (MTT), and area under the curve in percentage (AUC).

To qualitatively evaluate the intracranial pressure, ocular ultrasound is performed to measure the change of the optic nerve sheath diameter(mm). Elevation of intracranial pressure is considered if this diameter is above 0.55 mm

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with successful resuscitation after out-hospital or in-hospital cardiorespiratory arrest

Exclusion Criteria:

* Younger than 18 years old
* Pregnancy
* Acute or history of neurological disorder: stroke, bleeding, trauma, post-neurosurgery, tumor, meningitis.
* Severe dementia, psychiatric or neuromuscular disability
* Untreated Acute coronary syndrome
* Acute Respiratory Distress Syndrome (ARDS) with the ratio of arterial oxygen partial pressure (mmHg) to fractional inspired oxygen (PaO2/ FiO2) less than 150
* Severe systolic pulmonary hypertension above 90 mmHg
* Advanced liver cirrhosis with hyperammonemia
* Uremia > 200mmol/L
* Acute drug intoxications with coma
* Acute alcohol intoxication or withdrawal syndrome.
* Advanced malign diseases.
* History of allergy to the microbubble contrast SONOVUE.
* Insufficient echogenicity to ultrasound and incomplete insonation of the intracerebral arteries and brain parenchyma.
* Significant intracerebral and extracerebral arteries stenosis (≥ 70%) or vertebral artery hypoplasia (3mm).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change of the Mean transit time from baseline (seconds) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative evaluation of brain microcirculation using the variables of the time-intensity curve after Sonovue administration: a prolonged of Mean transit time is expected in comatose patients or non-survivors.
Mean change of the Peak intensity from baseline (dB). | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative evaluation of brain microcirculation using the variables of the time-intensity curve after Sonovue administration: a reduction of Peak intensity is expected in comatose patients or non-survivors.
Mean change of the time to Peak intensity from baseline (seconds). | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative evaluation of brain microcirculation using the variables of the time-intensity curve after Sonovue administration: a reduction of the time to peak intensity is expected in comatose patients or non-survivors.
Mean change of the Area under the curve from baseline (percentage). | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative evaluation of brain microcirculation using the variables of the time-intensity curve after Sonovue administration: a reduction of the area under the curve is expected in comatose patients or non-survivors.
Testing cerebral autoregulation: Transient Hyperemic test- Absence or presence from baseline | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Absence of cerebral autoregulation is considered if there is no change in flow velocities of the middle cerebral arteries after short compression of the common carotid arteries occur comparing with the value prior to compression.
Mean change of the optic nerve sheath diameter from baseline (mm) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative estimation of intracranial pressure using ocular ultrasound to measure the optic nerve sheath diameter. Elevation of intracranial pressure with increase of this diameter above 0.55 mm is expected in comatose patients or non-survivors.

SECONDARY OUTCOMES:
Mean change of the mean velocities of the middle cerebral arteries from baseline (cm/second) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative evaluation of brain macrocirculation using brain ultrasound to measure the velocities of the middle cerebral arteries. Unchanged or elevation of these velocities are expected in comatose patients or non-survivors.
Mean change of global cerebral blood flow from baseline (L/minute) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative evaluation of brain macrocirculation: using extracranial echo-color duplex to measure the velocities of both carotid and vertebral arteries to estimate global cerebral blood flow. Unchanged or elevation of cerebral blood flow is expected in comatose patients or non-survivors.
Mean change of cardiac output from baseline (L/minute) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 hours and at 72 or 96 hours
  Qualitative evaluation of brain macrocirculation: using transthoracic echocardiography to estimate cardiac output. Unchanged or elevation of cardiac output is expected in comatose patients or non-survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Duc Nam Nguyen, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robba C, Goffi A, Geeraerts T, Cardim D, Via G, Czosnyka M, Park S, Sarwal A, Padayachy L, Rasulo F, Citerio G. Brain ultrasonography: methodology, basic and advanced principles and clinical applications. A narrative review. Intensive Care Med. 2019 Jul;45(7):913-927. doi: 10.1007/s00134-019-05610-4. Epub 2019 Apr 25. PMID 31025061
- [Background] Piscaglia F, Nolsoe C, Dietrich CF, Cosgrove DO, Gilja OH, Bachmann Nielsen M, Albrecht T, Barozzi L, Bertolotto M, Catalano O, Claudon M, Clevert DA, Correas JM, D'Onofrio M, Drudi FM, Eyding J, Giovannini M, Hocke M, Ignee A, Jung EM, Klauser AS, Lassau N, Leen E, Mathis G, Saftoiu A, Seidel G, Sidhu PS, ter Haar G, Timmerman D, Weskott HP. The EFSUMB Guidelines and Recommendations on the Clinical Practice of Contrast Enhanced Ultrasound (CEUS): update 2011 on non-hepatic applications. Ultraschall Med. 2012 Feb;33(1):33-59. doi: 10.1055/s-0031-1281676. Epub 2011 Aug 26. No abstract available. PMID 21874631
- [Background] Harrois A, Duranteau J. Contrast-enhanced ultrasound: a new vision of microcirculation in the intensive care unit. Crit Care. 2013 Aug 23;17(4):449. doi: 10.1186/cc12860. PMID 24103639
- [Background] Seidel G, Meairs S. Ultrasound contrast agents in ischemic stroke. Cerebrovasc Dis. 2009;27 Suppl 2:25-39. doi: 10.1159/000203124. Epub 2009 Apr 16. PMID 19372658
- [Background] Geeraerts T, Merceron S, Benhamou D, Vigue B, Duranteau J. Non-invasive assessment of intracranial pressure using ocular sonography in neurocritical care patients. Intensive Care Med. 2008 Nov;34(11):2062-7. doi: 10.1007/s00134-008-1149-x. Epub 2008 May 29. PMID 18509619